CLINICAL TRIAL: NCT07048327
Title: Cohort Study of Intrauterine Diseases
Acronym: TJ Intrauterin
Status: Recruiting | Type: Observational
Sponsor: Wenwen Wang (Other)
Responsible Party: Sponsor-Investigator, Wenwen Wang, Clinical Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: CSID
Record Dates: First submitted 2025-06-19; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Endometrial Cancer; Endometrial Hyperplasia; Endometrial Polyps
Keywords: Intrauterine diseases; Endometrial Cancer; Endometrial Hyperplasia; Endometrial Polyps; Cohort Study
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intrauterine Diseases Cohort: Disease-specific cohort for uterine cavity diseases
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
"This study employs a prospective cohort design by establishing a uterine cavity diseases research platform. The investigators will collect participants' current medical history, menstrual and obstetric history, past medical history, physical and gynecological examinations, imaging studies, laboratory tests, and pathological examinations. After the hysteroscopic surgery, the investigators will conduct a one-year follow-up on the disease progression of the participants. Through this comprehensive approach, the investigators aim to deeply investigate the pathogenesis, risk factors, and optimized treatment strategies for uterine cavity diseases."

DETAILED DESCRIPTION:
Uterine cavity diseases are a common category of hormone-dependent gynecological conditions, encompassing a wide spectrum from benign lesions to malignant tumors, including endometrial hyperplasia, endometrial polyps, and endometrial malignancies.

Endometrial hyperplasia is classified into two types: hyperplasia without atypia and atypical hyperplasia. Atypical hyperplasia is considered a precancerous lesion of endometrial malignancies, which may lead to irregular vaginal bleeding, menstrual disorders, and carries the risk of malignant transformation. Endometrial polyps, a common benign lesion within the uterine cavity, often cause abnormal uterine bleeding, infertility, or recurrent miscarriages, significantly impacting women's reproductive health and quality of life. Endometrial malignancies, the most prevalent malignant tumors in the female reproductive system, pose a serious threat to women's lives and safety. These diseases not only profoundly affect women's physical health but also have far-reaching negative consequences on their mental well-being, social functioning, and overall quality of life.

In light of this, this study aims to utilize patients' clinical data resources to establish a cohort research platform for uterine cavity diseases, bridging the gap between clinical practice and scientific research, and providing valuable clinical data resources for in-depth studies on these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years;
* Patients requiring hysteroscopy or diagnostic curettage for intrauterine pathologies (e.g., endometrial hyperplasia, endometrial polyps, submucosal uterine fibroids, adenomyosis, or endometrial malignancies);
* Willing and able to comply with follow-up requirements;
* Signed informed consent obtained.

Exclusion Criteria:

* Concurrent participation in other drug clinical trials;
* Contraindications to or inability to tolerate hysteroscopy/curettage procedures;
* Unwilling or unable to provide informed consent;
* Unwilling or unable to adhere to study protocols.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population will be enrolled by a multicenter study led by Tongji Hospital , in collaboration with over 30 tertiary hospitals. Patients requiring hysteroscopic or curettage procedures for intrauterine lesions such as endometrial hyperplasia, polyps, and malignancies will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
The recurrence of endometrial polyps or endometrial hyperplasia. | Follow up every three months for one year after hysteroscopic surgery
  To evaluate the presence of disease progression and recurrence through imaging results.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared due to ethical restrictions and participant privacy protections outlined in the informed consent documents.